CLINICAL TRIAL: NCT00822575
Title: Relief From Itching of Mosquito Bites Clinical Study Protocol.
Brief Title: Study of a Device to Relieve Mosquito Bite Itching.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ecobrands, Ltd. (Industry)
Responsible Party: Mr. Robin Baker, EcoBrands, Ltd.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZC-001
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Mosquito Bites
Keywords: mosquito bites; itching
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Device: ZapperClick
- B (Sham Comparator)
  Interventions: Device: ZapperClick

INTERVENTIONS:
Device: ZapperClick — The ZapperClick is a therapeutic device that employs the piezo-electricity principle to soothe itching and ease the swelling from mosquito and horsefly bites as well as jellyfish and nettle stings. It accomplishes this by discharging 13KV at 0.7mA for 10 microseconds over the area of the bite or sting each time it is activated.

SUMMARY:
The purpose of this study is to determine whether over-the-counter (OTC) use of the ZapperClick device employing the piezo-electricity principle is effective in reducing itching associated with mosquito bites.

DETAILED DESCRIPTION:
The ZapperClick is a therapeutic device that employs the piezo-electricity principle to soothe itching and ease the swelling from mosquito and horsefly bites as well as jellyfish and nettle stings. It accomplishes this by discharging 13KV at 0.7mA for 10 microseconds over the area of the bite or sting each time it is activated. In this clinical study, only the indication of reducing itching from mosquito bites will be evaluated. The theory behind the device's effectiveness is that multiple high voltage, low current electrical discharges over a bug bite or sting generates warmth over the immediate area of the bite or sting which inhibits the histamine release, thus relieving the symptoms of itching and swelling arising from the bite or sting. The device is a quick, simple and painless means of reducing the annoying symptoms of mosquito bites.

ELIGIBILITY:
Inclusion Criteria:

* One lab-induced mosquito bite on the non-dominant forearm
* Familiarity with an immediate mosquito bite reaction.
* History of immediately responding to mosquito bites with itching.
* Willing and able to refrain from consuming anti-histamines, corticosteroids, or Non-Steroid Anti-Inflammatory Drugs (NSAID,) for a time period of 4 half lives of the drug prior to the beginning of the study, and continuing throughout the course of the study.
* Willing to abstain from the use of insect repellant and/or any treatment other than the test device for the relief of mosquito bite symptoms until after the study.
* Primary written and spoken language is English.

Exclusion Criteria:

* No history of prior affliction with mosquito bites.
* History of lack of reaction to mosquito and/or other insect bites that includes itching.
* History of hypersensitivity to the bites or stings of mosquitoes, bees or wasps.
* Presence of mosquito bites or other types of insect bite/stings on any location on the body.
* Current use of steroids.
* Use of insect repellants during the week prior to study start.
* Use of topical agents on the arm during the week prior to study start.
* Pacemaker, ICD or other implantable heart device.
* Therapeutic use of any type of electrical stimulation.
* Epilepsy.
* Diabetes.
* Presence of neurological disorder.
* Prior surgery to the forearm area.
* Infection or wound in the forearm area.
* Any skin or other disease or illness that can cause or influence skin itching, such as Psoriasis.
* Developmental disability or cognitive impairment that impacts the ability to read and/or to understand the content of the informed consent form or the device labeling and/or impacts the ability to read and/or to understand and/or to complete the study case report forms.
* Significant psychological disorder(s) for which treatment has become necessary, including anxiety and depression; psychiatric hospitalization.
* Pregnancy or lactation.
* Involvement in litigation and/or receiving disability benefits related to any kind of disability, injury, or other medical problem.
* Participation in research over the preceding 90 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change in degree of itching rating on a 0-100 VAS. | 10 minutes

SECONDARY OUTCOMES:
Changes in 0-100 VAS itching ratings, and changes in total area of mosquito bite erythema, across the 24-hour evaluation period. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Hill, Ph.D., Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Department of Infectious & Tropical Diseases, London School of Hygiene & Tropical Medicine,, London, United Kingdom